CLINICAL TRIAL: NCT06034925
Title: Randomized Controlled Trial Comparing the Tolerability and Efficacy of Maribavir vs. Valganciclovir for CMV Prophylaxis in High-Risk Kidney Transplant Recipients
Brief Title: Maribavir vs. Valganciclovir for CMV Prophylaxis in High-Risk Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, David J. Taber, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00125967
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Transplant Complication; CMV
MeSH Terms: interventions — maribavir; Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): valganciclovir 900mg once daily
  Interventions: Drug: Valganciclovir
- Intervention (Experimental): maribavir 400mg twice daily
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir — maribavir 400mg twice daily
  Arms: Intervention
Drug: Valganciclovir — valganciclovir 900mg once daily
  Arms: Control

SUMMARY:
The purpose of this study is to find out if there is a difference in how well the standard MUSC cytomegalovirus (CMV) prevention medicine works, compared to a different medicine, in preventing CMV infections in kidney transplant recipients who are at risk for this type of infection, while also assessing the tolerability of these two regimens. The two medication regimens being compared are Valganciclovir (FDA approved to prevent and treat CMV infection) vs Maribavir (FDA approved to treat CMV infection) plus Acyclovir (FDA approved to prevent HSV infection).

DETAILED DESCRIPTION:
Maribavir has been evaluated for the prevention of CMV infection in Phase II and Phase III trials within allogeneic stem cell transplant recipients. At 6-months post-transplant, the rates of CMV infection using PCR were not different between treatment and placebo arms, although the rates of pp65 antigenemia were lower in the Maribavir group. However, these studies used a low dose of 100mg PO BID. In subsequent studies within solid organ transplantation, Maribavir dosed at 400 to 1200mg PO BID was equally efficacious to valganciclovir for the treatment of CMV infection. Of note and importance to this proposal, the rates of neutropenia were 4-5% in the Maribavir treated patients vs. 15-18% in Valganciclovir patients. Thus, at an appropriate dose, Maribavir appears to have similar efficacy to Valganciclovir in treating CMV infection with a significantly reduced incidence of neutropenia. Currently, there is a lack of randomized controlled trials assessing the safety and efficacy of adequately dosed (=400mg PO BID) Maribavir for the prevention of CMV infection in solid organ transplant recipients.

Aim 1. Assess the incidence of leukopenia in those randomized to Maribavir vs. Valganciclovir prophylaxis in adult kidney transplant recipients at high-risk of CMV infection.

Hypothesis 1. The incidence of clinically meaningful leukopenia, defined as a WBC count of < 3,000 cells/mm3 and a reduction in total mycophenolate dose below 1,500 mg/day or valganciclovir dose below 900mg per day (adjusted for renal function), will be significantly lower in the Maribavir arm, as compared to the Valganciclovir arm.

Aim 2. Assess the efficacy of Maribavir vs. Valganciclovir prophylaxis in adult kidney transplant recipients at high-risk of CMV infection.

Hypothesis 2. The incidence of CMV infection and disease will be similar between the Maribavir arm, as compared to the Valganciclovir arm, at 3-, 6-, and 12-months post-transplant.

Aim 3. Assess the impact of Maribavir vs. Valganciclovir prophylaxis on healthcare utilization and costs in adult kidney transplant recipients at high-risk of CMV infection.

Hypothesis 3. Healthcare utilization will be lower in the Maribavir arm, as compared to the Valganciclovir arm, at 6- and 12-months post-transplant, driven predominantly by reduced number of telephone calls, televisits, and laboratory monitoring encounters.

Exploratory Aim 4. Assess the impact of Maribavir vs. Valganciclovir prophylaxis in adult kidney transplant recipients at high-risk of CMV infection on patient-reported outcomes for quality of life and satisfaction.

Exploratory Aim 5. Assess any differences in leukopenia, efficacy, healthcare utilization and patient reported outcomes by race and sex in patients randomized to Maribavir vs. Valganciclovir prophylaxis in adult kidney transplant recipients at high-risk of CMV infection.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient at study institution
* =7 days of transplant
* Received at least one dose of rATG induction or patient is D+/R- CMV serostatus

Exclusion Criteria:

* Age <18 years at time of transplant
* Recipient of pancreas, liver, heart, lung transplant
* Recipient of investigational, non-FDA approved medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of patients that develop leukopenia in those randomized to maribavir versus those randomized to valganciclovir prophylaxis in adult kidney transplant recipients at high-risk of CMV infection. | One year following transplant
  Leukopenia is defined as a white blood cell count <3000 cells/mm3
Compare the proportion of patients that develop cytomegalovirus (CMV) infection in those randomized to maribavir versus those randomized to valganciclovir prophylaxis in adult kidney transplant recipients at high-risk of CMV infection. | One year following transplant
  CMV infection is defined as having at least one CMV DNA PCR test of >1000 copies/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Culpepper H, Overstreet M, Soliman K, Casey M, Rice T, Lively K, Scalea J, McGillicuddy J, Patel N, Taber D. A Randomized Controlled Trial Comparing the Tolerability and Efficacy of Maribavir vs. Valganciclovir for Cytomegalovirus (CMV) Prophylaxis in High-Risk Kidney Transplant Recipients: Study Protocol. Cureus. 2025 Aug 27;17(8):e91110. doi: 10.7759/cureus.91110. eCollection 2025 Aug. PMID 41018408